CLINICAL TRIAL: NCT02422277
Title: Role of Low-intensity Shock Wave Therapy in Penile Rehabilitation Post Nerve Sparing Radical Cysto-prostatectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Zewin, Clinical Fellow in Urology and Nephrology center, Faculty of Medicine, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TZewin132015
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Bladder Cancer
Keywords: Cystoprostatectomy; Sexual function; Phosphodiestrase 5 inhibitors; Low intensity extracorporeal shock wave therapy; Erectile dysfunction; Penile rehabilitation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LI-ESWT group (Active Comparator): Intervention include that patients will undergo penile low-intensity extracorporeal shock wave therapy, 6-12 sessions, 1500 shocks per session, two sesssions per week for 3 weeks then 3 weeks break and then 2 sessions per week for 3 weeks.
  Interventions: Device: LI-ESWT group
- PDE-5 inhibitors group (Active Comparator): Intervention include that patients will intke oral tablets of PDE-5 inhibitors :
  - Oral intake of 50 mg once daily for 6 months.
  Interventions: Drug: PDE-5 inhibitors group
- Control group (No Intervention): Patients will be only followed up without any therapy for assisting erection.

INTERVENTIONS:
Device: LI-ESWT group — The patients in this arm will be subjected to Penile LI-SWT in the following parameters: 6 to 12 sessions with 1500 shocks per session. Each session will comprise the application of 300 shock waves (energy intensity of 0.09 mJ/mm2) to each of five different sites on the penis: three along the penile shaft and two at the crura with Frequency: 4 HZ. Energy level: 8 mJ/mm2. Rate: 120 shocks per minute.
  -Intervals: 2 treatment sessions per week for 3 weeks, then 3-weeks no-treatment interval, then 3-weeks treatment period of 2 treatment sessions per week.
  Other Names: shock wave group
  Arms: LI-ESWT group
Drug: PDE-5 inhibitors group — The patient in this arm will receive 50 mg of phosphodiesterase-5 inhibitors, oral intake once daily for 6 monthes.
  Other Names: Sildenafil
  Arms: PDE-5 inhibitors group

SUMMARY:
The aim of this clinical trial is to evaluate the role of extracorporeal low-intensity shock wave therapy in penile rehabilitation post nerve sparing radical cysto-prostatectomy.

DETAILED DESCRIPTION:
60 patients for whom nerve sparing radical cystoprostatectomy will be carrried out, penile rehabilitation by using low intensity extracorporeal shock wave therapy will be applied in 20 patients, another 20 patients will receive oral phosphodiestrase type 5 inhibitorrs and 20 patients will not receive any interventions in the control group.

ELIGIBILITY:
Inclusion Criteria:

- Patients will be eligible if he is sexually motivated and potent men with stable relationship of more than 6 months duration who will undergo nerve sparing radical cysto-prostatectomy for organ-confined bladder cancer.

Exclusion Criteria:

- 1. Men with Peyronie's disease. 2. Inflammation in the shock wave area. 3. Evidence of disease failure after surgery. 4. Patients developing postoperative complications requiring hospital readmission after surgery which interferes with the process of SWL.

5. Unstable medical or psychiatric disorder.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of sexual function by increase satisfaction and good vaginal penetration | 6 MOTHES
  increase in IIEF score by 5 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Asmy, MD, Study Director — a_assmy@yahoo.com
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt